CLINICAL TRIAL: NCT01882478
Title: CryoSpray Ablation for Barrett's Esophagus After Treatment Failure With Serial RadioFrequency Ablation
Brief Title: Cryotherapy -BEATS-RF Ablation Trial
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kenneth K. Wang, Kathy and Russ VanCleve Professor of Gastroenterology Reserach, Mayo Clinic
Other Study IDs: 12-006030
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Barrett's Esophagus With Persistent Dysplasia or; Early Esophageal Adenocarcinoma Post Radio Frequency Ablation
Keywords: Barrett's esophagus; Early esophageal adenocarcinoma; Radio Frequency Ablation; Cryotherapy
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- failure to respond to RF ablation: patients undergoing endoscopic RF ablation therapy with persistent BE with HGD or IMCA despite 2 or more serial RF ablation treatment sessions

SUMMARY:
The purpose of this study is to determine whether cryotherapy is effective in the treatment of persistent high grade dysplasia (HGD) or early esophageal adenocarcinoma (IMCA) in patients who have not responded to radiofrequency ablation (RFA).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Able to provide informed consent
* Patients with unifocal or multifocal BE with HGD or IMCA who have failed at least 2 serial RFA therapy.
* Patients who refused esophagectomy or deemed inoperable or whose BE dysplasia is not amenable to endoscopic mucosal resection (EMR) treatment alone due to: (1) extensive multifocal lesions (2) severe coagulopathy or any medical condition deemed high risk for EMR (3) patient refuses EMR
* Patients with a nodular BE lesions may undergo clinically-indicated EMR and still be eligible for enrollment as long as they have BE-HGD lesion/s that are still candidate for ablative treatment

Exclusion Criteria:

* Age younger than 18 years old
* Life expectancy less than 12 months
* Pregnancy
* Presence of esophageal varices
* Esophageal stricture precluding passage of an endoscope and suction tubing
* Any procedure that has impeded normal gastric emptying or limited gastric volume distention, including but not limited to gastric bypass, stomach stapling, gastrojejunostomy or any disease state has significantly reduced the elasticity in the GI tract (e.g. Marfan's syndrome, Scleroderma or any Connective Tissue Disease)
* Esophageal cancer (T2 and above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with persistent BE with HGD or IMCA despite 2 or more serial RF ablation treatment sessions in a cohort of patients undergoing endoscopic therapy.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-06; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Response | 2 years
  To assess efficacy of achieving elimination of dysplasia in patients with RFA-refractory BE with HGD or IMCA

SECONDARY OUTCOMES:
Predictors of response | 2 years
  To identify potential predictors of CE-D and CE-IM in patients requiring rescue CSA treatment after failed RFA therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth K Wang, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials